CLINICAL TRIAL: NCT00988325
Title: An Open Label, Prospective, Pharmacokinetic/Pharmacodynamic and Safety Evaluation of Oseltamivir (Tamiflu®) in the Treatment of Infants 0 to <12 Months of Age With Confirmed Influenza Infection
Brief Title: A Pharmacokinetic/Pharmacodynamic (PK/PD) and Safety Evaluation of Oseltamivir [Tamiflu] in the Treatment of Infants 0 to <12 Months of Age With Confirmed Flu Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WP22849; 2009-014365-12
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

ARMS (3):
- Oseltamivir 3 mg (Experimental): infants 3 to <12 months
  Interventions: Drug: Tamiflu
- Oseltamivir 2.5 mg (Experimental): infants 1 to <3 months of age
  Interventions: Drug: Tamiflu
- Oseltamivir 2 mg (Experimental): infants 0 to 30 days (post natal) of age
  Interventions: Drug: Tamiflu

INTERVENTIONS:
Drug: Tamiflu — oral repeating dose

SUMMARY:
This study will assess the pharmacokinetics/pharmacodynamics and safety of oseltamivir [Tamiflu] therapy in infants less than 1 year of age with influenza diagnosed in the 96 hours prior to the first dose. Patients age 3-12 months will receive 3 mg/kg, 1-3 months will receive 2.5 mg/kg, and birth to 1 month will receive 2 mg/kg twice a day for a total of 10 doses. Patients positive for influenza virus on Day 6 will be eligible to receive continued study treatment for an additional 10 doses (5 days). The anticipated time on study treatment is 4 weeks, and the target sample size is 65-85 male and female infants.

ELIGIBILITY:
Inclusion Criteria:

* infants </=12 months of age
* laboratory confirmed diagnosis of influenza within 96 hours prior to first dose
* influenza symptoms for </=96 hours prior to first dose

Exclusion Criteria:

* preterm infants less than 40 weeks (corrected for gestational age)
* weight less than 5th percentile for age (corrected for gestational age)
* concurrent gastrointestinal conditions that preclude enteric absorption of the drug
* bronchopulmonary dysplasia/chronic lung disease on assisted ventilation at time of enrollment
* active or uncontrolled respiratory, cardiac, hepatic, CNS or renal disease at baseline
* symptomatic inborn errors of metabolism

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Cliniques Universitaires St-Luc, Brussels, Belgium
- Hôpital Femme Mère Enfant; Service de rhumatologie pédiatrique, Bron, France
- Germany (3):
  - CAMPUS VIRCHOW-KLINIKUM CharitéCentrum 17 Klinik f.Pädiatrie Abt.Pneumologie u.Immunologie, Berlin
  - LWL-Klinik-Bochum, Bochum
  - Onkologische Schwerpunktpraxis Dr. Med. O. Burkhard & B. Reimann, Worms
- Fondazione Ospedale Maggiore Policlinico, Milan, Lombardy, Italy
- Poland (4):
  - Vitamed, Bydgoszcz
  - Samodzielny Publiczny Zakład Opieki; Wcześniaków I Intensywnej Terapii, Bydgoszcz
  - Zespol Opieki Zdrowotnej Debica; Oddzial Dzieciecy, Dębica
  - St Hedwig Hospital In Trzebnica, Trzebnica
- Spain (2):
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Intermedios y Urgencias Pediatricas, Santiago de Compostela, La Coruña
  - Hospital Universitario de Getafe; Servicio de Pediatria, Madrid, Madrid

REFERENCES:
- [Derived] Rath BA, Brzostek J, Guillen S, Niranjan V, Chappey C, Rayner CR, Clinch B. Safety, virology and pharmacokinetics of oseltamivir in infants with laboratory-confirmed influenza: a Phase I/II, prospective, open-label, multicentre clinical trial. Antivir Ther. 2015;20(8):815-25. doi: 10.3851/IMP2967. Epub 2015 May 27. PMID 26015411

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 11 centers in Spain, Italy, France, Germany, Belgium, and Poland from 10 January 2011 to 04 April 2012. A total of 65 participants were screened.
Groups:
- Oseltamivir 3 mg/kg: Participants aged 91 to <365 days received oral suspension of oseltamivir 3 milligram (mg)/kilogram (kg) twice a day for 5 days
- Oseltamivir 2.5 mg/kg: Participants of age 31 to 90 days received oral suspension of oseltamivir 2.5 mg/kg twice a day for 5 days
- Oseltamivir 2 mg/kg: Participants of age 0 to 30 days received oral suspension of oseltamivir 2 mg/kg twice a day for 5 days.
Period: Overall Study
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Started | 40 | 20 | 5
Completed | 40 | 20 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all treated participants with at least one post-baseline safety assessment (vital sings like temperature, respiratory rate, blood pressure, pulse rate).
Groups:
- Oseltamivir 3 mg/kg: Participants aged 91 to <365 days received oral suspension of oseltamivir 3 mg/kg twice a day for 5 days.
- Total: Total of all reporting groups
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg | Total
Number analyzed (Participants) | 40 | 20 | 5 | 65
Age, Continuous [Mean (Standard Deviation); unit: Days] | 223.2 (79.41) | 57.0 (17.24) | 25.2 (5.36) | 156.8 (105.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 8 | 2 | 29
  Male | 21 | 12 | 3 | 36

OUTCOME MEASURES:

1. Primary Outcome: Steady-state Area Under the Plasma Concentration Versus Time Curve From Time Zero to 12 Hours of Oseltamivir and Oseltamivir Carboxylate
Description: Oseltamivir carboxylate is active metabolite of oseltamivir. AUC0-12 was estimated for oseltamivir and oseltamivir carboxylate by linear trapezoidal rule
Time Frame: 15 minutes pre-dose; 1 hour +/- 15 minutes, 2-3, 5-7, 10-12 hours post-dose on Day 3 if two doses taken on Day 1 or 15 minutes pre-dose; 1 hour +/- 15 minutes, 2-3, 5-7, 10-12 hours post-dose on Day 4 if one dose taken on Day 1
Population: Pharmacokinetic (PK) population included all treated participants with at least one blood sample evaluable for drug concentration level and who adhered to the protocol. n = participants with evaluable drug concentration
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)*nanogram(ng)/milliliter (mL)
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 40 | 20 | 5
hour (h)*nanogram(ng)/milliliter (mL)
  Oseltamivir, n=37, 17, 4 | 277 (36.2) | 194 (47.8) | 142 (48.8)
  Oseltamivir carboxylate, n=18,11, 2 | 4990 (27.4) | 4920 (35.3) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated for 2 participants analyzed. Individual data are not reported due to privacy concerns

2. Secondary Outcome: Time to the Maximum Observed Plasma Concentration of Oseltamivir and Oseltamivir Carboxylate
Description: Oseltamivir carboxylate is an active metabolite of oseltamivir.Tmax was estimated using non-compartmental methods
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 40 | 20 | 5
hours
  Oseltamivir | 1.08 [0.88 to 3.08] | 1.08 [0.00 to 2.92] | 1.08 [1.00 to 3.00]
  Oseltamivir carboxylate | 5.04 [2.08 to 7.00] | 2.88 [0.00 to 6.67] | 5.83 [2.58 to 6.67]

3. Secondary Outcome: Apparent Elimination Half Life of Oseltamivir and Oseltamivir Carboxylate
Description: Elimination half-life is defined as the time required for elimination of a drug to half its plasma concentration and was computed using non-compartmental method
Time Frame: 15 minutes pre-dose; 1 hour +/- 15 minutes, 2-3, 5-7, 10-12 hours post-dose on Day 3 if two doses taken on Day 1 or 15 minutes pre-dose; 1 hour +/-15 minutes, 2-3, 5-7, 10-12 hours post-dose on Day 4 if one dose taken on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 40 | 20 | 5
hours
  Oseltamivir, n= 37, 17, 4 | 2.02 (38.5) | 2.01 (49.3) | 1.66 (41.5)
  Oseltamivir carboxylate, n=18, 11, 2 | 9.45 (53.3) | 11.3 (92.7) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated for 2 participants analyzed. Individual data are not reported due to privacy concerns

4. Secondary Outcome: Apparent First-order Elimination Rate Constant of Oseltamivir and Oseltamivir Carboxylate
Description: Oseltamivir carboxylate is active metabolite of oseltamivir.The apparent first-order elimination rate constant (Lambda Z) was determined by linear regression analysis of terminal data points. A minimum of 3 data points were used for lambda Z estimation. By reporting tool convention, if n<3, no summary statistics were calculated
Time Frame: as for outcome 1
Population: Pharmacokinetic (PK) population included all treated participants with at least one blood sample evaluable for drug concentration level and who adhered to the protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 40 | 20 | 5
1/hour
  Oseltamivir, n= 33, 11, 4 | 0.349 (39.9) | 0.338 (52.9) | 0.418 (41.5)
  Oseltamivir carboxylate, n=17, 7, 2 | 0.0735 (55.2) | 0.0475 (110.6) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated for 2 participants analyzed. Individual data are not reported due to privacy concerns

5. Primary Outcome: Steady-state Maximum Observed Plasma Concentration of Oseltamivir and Oseltamivir Carboxylate
Description: Oseltamivir carboxylate is an active metabolite of oseltamivir. Cmax was estimated for both oseltamivir and Oseltamivir carboxylate by non-compartmental analysis.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 40 | 20 | 5
ng/mL
  Oseltamivir | 80.8 (47) | 62.5 (69.1) | 25.2 (211.6)
  Oseltamivir carboxylate | 464 (37.7) | 530 (33.1) | 501 (22.2)

6. Primary Outcome: Steady-state Minimum Observed Plasma Concentration of Oseltamivir and Oseltamivir Carboxylate
Description: Oseltamivir carboxylate is active metabolite of oseltamivir. Cmin was estimated for both oseltamivir and oseltamivir carboxylate by non-compartmental analysis
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 40 | 20 | 5
ng/mL
  Oseltamivir | 2.88 (65.4) | 2.09 (52.6) | 2.56 (90.0)
  Oseltamivir carboxylate | 238 (43.8) | 248 (51.5) | 169 (96.4)

7. Secondary Outcome: Total Plasma Clearance as a Function of Bioavailability and Apparent Plasma Clearance of the Metabolite as a Function of Bioavailability (CLm/F) of Oseltamivir and Oseltamivir Carboxylate
Description: Oseltamivir carboxylate is active metabolite of oseltamivir. CL/F was calculated as dose/AUCinf, where AUCinf represents the area under the concentration-time curve of the analyte in plasma over the time interval from zero extrapolated to infinity
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/hour
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 40 | 20 | 5
mL/hour
  Oseltamivir, n= 37, 17, 4 | 80500 (42.8) | 63000 (63.7) | 50600 (39.9)
  Oseltamivir carboxylate, n=18,11, 2 | 3940 (38.8) | 2180 (54.86) | NA (NA) — Total Plasma Clearance was not calculated for 2 participants analyzed. Individual data are not reported due to privacy concerns

8. Secondary Outcome: The Volume of Distribution as a Function of Bioavailability of Oseltamivir and Oseltamivir Carboxylate
Description: Oseltamivir carboxylate is active metabolite of oseltamivir. V/F is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 40 | 20 | 5
mL
  Oseltamivir, n= 37, 17, 4 | 234000 (66.2) | 183000 (87.9) | 121000 (69.8)
  Oseltamivir carboxylate, n=18,11, 2 | 53700 (78.1) | 35400 (96.5) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated for 2 participants analyzed. Individual data are not reported due to privacy concerns

9. Secondary Outcome: Clast of Oseltamivir and Oseltamivir Carboxylate
Description: The last measurable plasma concentration of oseltamivir and oseltamivir carboxylate was the last quantifiable concentration of oseltamivir or oseltamivir carboxylate, respectively.
Time Frame: as for outcome 1
Population: Pharmacokinetic (PK) population included all treated patients with at least one blood sample evaluable for drug concentration level and who were adhered to the protocol
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 40 | 20 | 5
ng/mL
  Oseltamivir | 262 (39.2) | 176 (58.3) | 84.3 (154.4)
  Oseltamivir carboxylate | 3800 (50.1) | 4410 (34.0) | 3940 (28.2)

10. Secondary Outcome: Time of the Last Measurable Plasma Concentration for Oseltamivir and Oseltamivir Carboxylate
Description: Oseltamivir carboxylate is an active metabolite of oseltamivir.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 40 | 20 | 5
hours
  Oseltamivir | 9.23 (30.1) | 8.53 (32.9) | 6.94 (24.2)
  Oseltamivir carboxylate | 10.11 (21.2) | 10.64 (5.4) | 10.45 (5.3)

11. Secondary Outcome: Number of Participants With Change From Baseline in Neurological Assessment Scores
Description: Neurological assessment was performed to assess the mental state of the participants through two scales: Infant face scale and Glasgow coma scale. Each scale consists of 3 subscales: eye opening (ranging 1 to 4), verbal response (ranging 1 to 5), and motor responses (ranging 1 to 6). The final score is the sum of these ranges and is scored between 3 and 15. 3 being the worst, and 15 the best. Change from baseline is change of final score post-baseline minus the final score at baseline.
Time Frame: Baseline (Day 1); Day 3 for who received two does on Day 1 or Day 4 for who received one dose on Day 1; Day 6, Day 11, Day 18, Day 30
Population: Safety population included all treated participants with at least one post-baseline safety assessment
Measure: Number; unit: participants
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 40 | 20 | 5
participants
  With change in infant face scale measurement score | 0 | 2 | 0
  With change in Glasgow coma scale assessment score | 0 | 1 | 0

12. Secondary Outcome: Median Time to Cessation of Viral Shedding in Participants With Positive Culture at Baseline
Description: Median time to cessation of viral shedding was calculated for all patients with positive by culture / by polymerase chain reaction (PCR) at baseline using all data points between the start of the treatment and the 1st time point of negative culture without subsequent positive culture results. These time-to event analyses were only performed for the viral titre.
Time Frame: Days 1, 3 or 4, 6, 11, 18, and 30
Population: Pharmacodynamic Analysis Population consisted of all enrolled participants with a positive influenza infection confirmed by culture or PCR at baseline or anytime during the study
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 40 | 20 | 5
hours | 228.5 [118.0 to 231.0] | 113.0 [63.0 to 230.0] | 113.0 [110.0 to 116.0]
Statistical Analysis 1: Comparison: Oseltamivir 3 mg/kg vs Oseltamivir 2.5 mg/kg vs Oseltamivir 2 mg/kg; Test type: Superiority or Other; p = 0.166, Wilcoxon (Mann-Whitney) — p-value is for the comparison of the age cohorts (treatment groups); Wilcoxon Test was used for testing homogeneity of survival curves; Median time to cessation of viral sheddi = 119, 95% CI 2-sided [113 to 230] — Median time was estimated from the Kaplan-Meier curve (unstratified)

13. Secondary Outcome: Number of Participants With Virus Shedding by Virus Type
Description: The viral titer was measured by culture and reported in log10 (50% tissue culture infective dose [TCID50]). The viral load was analyzed by PCR and reported as log10 particles/mL. The number of patients positive for viral shedding by virus sub-type was measured on specified days from baseline to last visit on Day 30.
Time Frame: Baseline (Day 1), Day3/4, Day 6, Day 11, Day 18+/-2 days, Day 30+/-2 days
Population: as for outcome 12
Measure: Number; unit: Participants
Groups:
- Type A (H1N1)pdm09: Genotype A (H1N1)pdm09 was present in 21 participants of age group 91 to <365 days, 9 participants of age group 31 to 90 days, and 2 participants of age group <=30 days
- Type A H3: Genotype Type A H3 was present in 4 participants and 6 participants of age groups 91 to <365 days and 31 to 90 days, respectively
- Type B: Genotype B was present in 12, 2, and 2 participants of age groups <365 days, 31 to 90 days, and <=30 days, respectively.
Arm/Group | Type A (H1N1)pdm09 | Type A H3 | Type B
Number analyzed (Participants) | 32 | 10 | 16
Participants
  Baseline | 32 | 10 | 14
  Day 3 or 4 | 20 | 5 | 14
  Day 6 | 12 | 4 | 7
  Day 11 | 32 | 9 | 16
  Day 18 +-2 | 0 | 1 | 0
  Day 30 +-2 | 0 | 0 | 0

14. Secondary Outcome: Time to Resolution of Fever in Participants With Fever at the Baseline
Description: This was performed for all participants who had fever at baseline. Fever is defined as body temperature >37.0 degree Celsius. Rectal temperature is converted by subtracting 1 degree Celsius. Time to Resolution of Fever was defined as the time from the initiation of treatment to first time the afebrile state was reached and maintained for at least 21.5 hours, where afebrile state was defined as axillary temperature ≤ 37 degree Celsius.
Time Frame: Days 1 to 11; Day 18; Day 30
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 37 | 17 | 4
hours | 12.0 [9.0 to 17.0] | 20.5 [12.0 to 36.0] | 24.0 [14.0 to 43.0]
Statistical Analysis 1: Comparison: Oseltamivir 3 mg/kg vs Oseltamivir 2.5 mg/kg vs Oseltamivir 2 mg/kg; Test type: Superiority or Other; p = 0.059, Wilcoxon (Mann-Whitney) — The p-value is for the comparison of the age cohorts (not including Total); Time to Resolution of Fever in Patients = 14.5, 95% CI 2-sided [12 to 20] — Median time was estimated from the Kaplan-Meier curve (unstratified)

15. Secondary Outcome: Percentage of Participants With Decline of Body Temperature to the Afebrile State
Description: This was performed for all participants who had fever at baseline Fever is defined as body temperature >37.0ºC. Rectal temperature is converted by subtracting 1 ºC. The rate of decline of body temperature was calculated as the slope of body temperature between the baseline temperature and the 1st temperature below 37°C. Participants with decline in body temperature were considered to have no fever; however, participants who did not show any decline in body temperature were considered to have persisting fever.
Time Frame: Baseline (Day 1), Day3/4, Day 6, Day 11, Day 18+/-2 days, Day 30+/-2 days
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 33 | 11 | 4
percentage of participants
  Baseline, n=33, 11, 4, decline | 36 | 55 | 25
  Baseline, n=33, 11, 4, no decline | 64 | 45 | 75
  Day 4, n=33, 11, 4, decline | 94 | 91 | 100
  Day 4, n=33, 11, 4, no decline | 6 | 9 | 0
  Day 11, n=33, 11, 4, decline | 97 | 100 | 100
  Day 11, n=33, 11, 4, no decline | 3 | 0 | 0
  Day 18, n=16, 5, 1, decline | 94 | 100 | 100
  Day 18, n=16, 5, 1, no decline | 6 | 0 | 0
  Day 30, n=31, 9, 4, decline | 97 | 89 | 100
  Day 30, n=31, 9, 4, no decline | 3 | 11 | 0

16. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Secondary Illness
Description: An Adverse Event (AEs) is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An Serious Adverse Event (SAE) is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect. Secondary illnesses were influenza disease-related events, namely bronchitis, pneumonia, otitis media, and sinusitis that resolved without sequelae. Adverse events, serious adverse events, and secondary illness are reported for on-treatment period (from the first dose of oseltamivir upto 3 days after the last dose of oseltamivir [Approximately 14 days].
Time Frame: Up to 3 days after the last dose of oseltamivir (Approximately 14 days)
Population: Safety population included all treated participants with at least one post-baseline safety assessment
Measure: Number; unit: Participants
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 40 | 20 | 5
Participants
  Participants with any AE | 13 | 12 | 2
  Participants with any SAE | 3 | 1 | 0
  Participants with secondary illness | 0 | 1 | 0

17. Secondary Outcome: Number of Participants Showing Within-patient Variability in Vital Signs
Description: Systolic blood pressure, diastolic blood pressure, pulse rate, respiratory rate, and heart rate were examined for any consistent within-patient post-baseline changes.
Time Frame: Post baseline, Day 3, 4, 6, 11, 18+/- 2 days, 30+/-2 days
Population: Safety population included all treated participants with at least one post-baseline safety assessment. Due to the small numbers of participants and the extent of influenza induced variability, changes in vital sign patterns cannot be detected.
Arm/Group | Oseltamivir 3 mg/kg | Oseltamivir 2.5 mg/kg | Oseltamivir 2 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 days after the last dose of oseltamivir (Approximately 14 days)
Description: SAEs and other AEs were collected in the safety population. Safety population included all treated participants with at least one post-baseline safety assessment. All AEs are reported for on-treatment period (from the first dose of oseltamivir up to 3 days after the last dose of oseltamivir [Approximately 14 days].
Groups:
- Oseltamivir 3 mg: Participants aged 91 to <365 days received oral suspension of oseltamivir 3 milligram (mg)/kilogram (kg) twice a day for 5 days
- Oseltamivir 2.5 mg: Participants of age 31 to 90 days received oral suspension of oseltamivir 2.5 mg/ twice a day for 5 days
- Oseltamivir 2 mg: Participants of age 0 to 30 days received oral suspension of oseltamivir 2 mg/kg twice a day for 5 days
Arm/Group | Oseltamivir 3 mg | Oseltamivir 2.5 mg | Oseltamivir 2 mg
Serious Adverse Events (participants affected / at risk) | 3/40 | 1/20 | 0/5
Other Adverse Events (participants affected / at risk) | 13/40 | 12/20 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oseltamivir 3 mg (N=40) | Oseltamivir 2.5 mg (N=20) | Oseltamivir 2 mg (N=5)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 1 | 0
Cellulitis orbital (Infections and infestations) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oseltamivir 3 mg (N=40) | Oseltamivir 2.5 mg (N=20) | Oseltamivir 2 mg (N=5)
Vomiting (Gastrointestinal disorders) | 10 | 11 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 0
Regurgitation (Gastrointestinal disorders) | 1 | 6 | 2
Pyrexia (General disorders) | 3 | 0 | 0
Irritability (General disorders) | 0 | 2 | 0
Crepitations (General disorders) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 1
Rotavirus infection (Infections and infestations) | 1 | 1 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 2 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.